CLINICAL TRIAL: NCT05576974
Title: A Phase 2a, Single-dose, Open-label Study to Evaluate Diagnostic Performance and Safety of Pegsitacianine, an Intraoperative Fluorescence Imaging Agent for the Detection of Cancer, in Patients With Unknown Primary Head and Neck Cancer (ILLUMINATE STUDY)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Baran Sumer, Professor and Chief, Division of Head and Neck Oncology, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2022-0460; 1R01CA266146-01 (NIH)
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Cancer; Unknown Primary Cancer; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Unknown Primary; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: In Part 1 the single dose of 1 mg/kg of pegsitacianine given 6-300 hours prior to surgery will be used to image primary tumors in patients with HNSCC to evaluated to verify the diagnostic performance of pegsitacianine fluorescence imaging for detecting primary tumors and metastatic lymph nodes.
  In Part 2, pegsitacianine the single dose of 1 mg/kg of given 6-300 hours prior to surgery will be used to in patients with unknown primary cancer of the head and neck. These patients typically undergo exam under anesthesia with a laryngoscopy as well as panendoscopy for identifying the source of the metastatic cancer found in the cervical nodes. Subjects for Part 2 may begin dosing at any time during Part 1 thus the two parts can run concurrently.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 - Cohort A (Active Comparator): In Part 1 the single dose of 1 mg/kg of pegsitacianine given 6-300 hours prior to surgery will be used to image primary tumors in patients with HNSCC to evaluated to verify the diagnostic performance of pegsitacianine fluorescence imaging for detecting primary tumors and metastatic lymph nodes.
  Interventions: Drug: Pegsitacianine
- Part 2 - Cohort B (Active Comparator): In Part 2, pegsitacianine the single dose of 1 mg/kg of given 6-300 hours prior to surgery will be used to in patients with unknown primary cancer of the head and neck. These patients typically undergo exam under anesthesia with a laryngoscopy as well as panendoscopy for identifying the source of the metastatic cancer found in the cervical nodes. The diagnostic performance of pegsitacianine fluorescence imaging for detecting primary tumors and metastatic lymph nodes in these patients will be evaluated. All the available data to date will be used to decide the additional tumor type(s), number of patients per tumor type, and number of Group(s) to be enrolled.
  Interventions: Drug: Pegsitacianine

INTERVENTIONS:
Drug: Pegsitacianine — Infusion of the Pegsitacianine-Intraoperative fluorescence imaging

SUMMARY:
This is a non-randomized, open-label, single-center, safety and imaging feasibility study of Pegsitacianine, an intraoperative fluorescence imaging agent.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single-center, safety and imaging feasibility study of Pegsitacianine, an intraoperative fluorescence imaging agent.

The main purpose of this study is to investigate whether Pegsitacianine can be used to image head and neck cancers as well as unknown primary cancer of the head and neck 6-300 hours post dose in patients undergoing routine surgery for biopsy, evaluation, detection or removal of their primary cancer.

The study consists of two Parts.

* Part 1 will be performed in a single dose of 1 mg/kg given such that Pegsitacianine fluorescence can be used to image primary tumors in patients with HNSCC undergoing routine surgery at 6-300 hours, and if needed at an alternate imaging schedule post dose.
* Part 2 will be performed in a single dose of 1 mg/kg given such that Pegsitacianine fluorescence can be used to image primary tumors in patients with unknown primary cancer of the head and neck (UPC) at 6-300 hours, and if needed at an alternate imaging schedule post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age
2. Biopsy-confirmed diagnosis, for primary or recurrent disease (or high clinical suspicion in the opinion of the Investigator)

   1. Part 1: Stage 1 to 4 HNSCC
   2. Part 2: UPC squamous cell carcinoma of the head and neck with metastatic disease to at least a single cervical node, AND no biopsy proven evidence of the primary cancer's location.
3. Acceptable hematologic status (as standard surgery protocol requires, as determined by the Investigator), kidney function and liver function. Elevations of creatinine, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or total bilirubin >1.5× the upper limit of normal [ULN] must be determined to be not clinically significant by the Investigator and approved by the Medical Monitor.
4. Documented negative serum pregnancy test for women of childbearing potential (i.e., premenopausal women with intact reproductive organs and women <2 years after menopause)
5. Male patients and female patients of child-bearing potential (i.e., premenopausal women with intact reproductive organs and women <2 years after menopause) must agree to and comply with using medically acceptable contraception including surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, bilateral tubal ligation), intrauterine device, oral contraceptive, contraceptive patch, long acting injectable contraceptive, partner's vasectomy, double-barrier method (condom or diaphragm plus spermicide or condom plus diaphragm), or abstinence during the trial and for 6 months thereafter
6. Agree to abstain from alcohol consumption from 72 hours before Pegsitacianine administration through completion of Study Day 10 (±48 hours) visit in Part 1 and Part 2.
7. Adequate potential for follow up

Exclusion Criteria:

1. Tumors at sites of which the surgeon would assess that in vivo intraoperative imaging would not be feasible.
2. Life expectancy <12 weeks
3. Karnofsky Performance Status <70%
4. Hepatic impairment (Child-Pugh score >5) or significant liver disease including active hepatitis or cirrhosis
5. Lab values or any sign, symptom, or medical condition that in the opinion of the PI would prevent surgical resection
6. Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
7. Pregnant or lactating women
8. Receiving or planned to receive, during the duration of the study, concomitant medication with a high chance of hepatotoxicity, as judged by the PI based on standard protocols within the study center
9. Alcohol consumption within 72 hours before Pegsitacianine administration
10. Received an investigational agent within the shorter of 5 half-lives or 30 days before Pegsitacianine dosing
11. Inability to adhere to the schedule of assessments or any circumstance that would interfere with the validity of assessments performed in the study
12. The PI considers that the patient should not participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostics performance and safety of 1 mg/kg Pegsitacianine in patients with HNSCC | 5 years
  Pegsitacianine fluorescence from in vivo and excised tissues will be imaged using intraoperative and post-operative NIR cameras and will be correlated with the histopathological confirmation of tumor and normal tissues to determine Pegsitacianine's diagnostic performance. Patient safety will be assessed for 10 days (±48 hours) post dose. All patients will be monitored for vital signs and physical examination pretreatment and at various time points up to Day 6 (±24 hours). All patients will be monitored for comprehensive metabolic panel (CMP) and complete blood count (CBC) with differentials pretreatment and at various time points up to Day 10 (±48 hours). All patients will be monitored for TEAEs, and concomitant medication use from the start of dosing up to Day 10 (±48 hours). TEAEs will be followed closely during the study to identify any potential DLTs
Diagnostics performance and safety of 1 mg/kg Pegsitacianine in patients with UPC | 5 years
  Pegsitacianine fluorescence from in vivo and excised tissues will be imaged using intraoperative and post-operative NIR cameras and will be correlated with the histopathological confirmation of tumor and normal tissues to determine Pegsitacianine's diagnostic performance. Patient safety will be assessed for 10 days (±48 hours). All patients will be monitored for vital signs and physical examination pretreatment and at various time points up to Day 6 (±48 hours). All patients will be monitored for comprehensive metabolic panel (CMP) and complete blood count (CBC) with differentials pretreatment and at various time points up to Day 10 (±48 hours). All patients will be monitored for TEAEs, and concomitant medication use from the start of dosing up to Day 10 (±48 hours). TEAEs will be followed closely during the study to identify any potential DLTs

SECONDARY OUTCOMES:
Pegsitacianine fluorescence imaging in HNSCC, UPC primary cancers that are HPV positive and HPV negative | 5 years
  Pegsitacianine fluorescence from in vivo and excised tissues will be imaged using intraoperative and post-operative NIR cameras and will be correlated with the histopathological confirmation of tumor and normal tissues to determine Pegsitacianine's diagnostic performance. Assessment of use of Pegsitacianine for intra-operative imaging of HNSCC, UPC and metastatic lymph nodes will include quantification of intraoperative and postoperative fluorescence signals from histology confirmed tumor and normal tissues, calculation of TBR and diagnostic performance. Feasibility determination will be based on a combined assessment of intraoperative in vivo and ex vivo fluorescent signals together with ex vivo examinations (histological examination, NIR flatbed scanning).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amit M, Yen TC, Liao CT, Chaturvedi P, Agarwal JP, Kowalski LP, Kohler HF, Ebrahimi A, Clark JR, Cernea CR, Brandao JS, Kreppel M, Zoller JE, Leider-Trejo L, Bachar G, Shpitzer T, Bolzoni AV, Patel RP, Jonnalagadda S, Robbins TK, Shah JP, Patel SG, Gil Z. The origin of regional failure in oral cavity squamous cell carcinoma with pathologically negative neck metastases. JAMA Otolaryngol Head Neck Surg. 2014 Dec;140(12):1130-7. doi: 10.1001/jamaoto.2014.1539. PMID 25074731
- [Background] Dacosta RS, Wilson BC, Marcon NE. Spectroscopy and fluorescence in esophageal diseases. Best Pract Res Clin Gastroenterol. 2006 Feb;20(1):41-57. doi: 10.1016/j.bpg.2005.08.003. PMID 16473800
- [Background] Davies B, Morris T. Physiological parameters in laboratory animals and humans. Pharm Res. 1993 Jul;10(7):1093-5. doi: 10.1023/a:1018943613122. No abstract available. PMID 8378254
- [Background] Denaro N, Russi EG, Adamo V, Merlano MC. State-of-the-art and emerging treatment options in the management of head and neck cancer: news from 2013. Oncology. 2014;86(4):212-29. doi: 10.1159/000357712. Epub 2014 May 10. PMID 24820548
- [Background] d'Alessandro AF, Pinto FR, Lin CS, Kulcsar MA, Cernea CR, Brandao LG, Matos LL. Oral cavity squamous cell carcinoma: factors related to occult lymph node metastasis. Braz J Otorhinolaryngol. 2015 May-Jun;81(3):248-54. doi: 10.1016/j.bjorl.2015.03.004. Epub 2015 Mar 30. PMID 25890681
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Gioux S, Choi HS, Frangioni JV. Image-guided surgery using invisible near-infrared light: fundamentals of clinical translation. Mol Imaging. 2010 Oct;9(5):237-55. PMID 20868625
- [Background] Haka AS, Volynskaya Z, Gardecki JA, Nazemi J, Lyons J, Hicks D, Fitzmaurice M, Dasari RR, Crowe JP, Feld MS. In vivo margin assessment during partial mastectomy breast surgery using raman spectroscopy. Cancer Res. 2006 Mar 15;66(6):3317-22. doi: 10.1158/0008-5472.CAN-05-2815. PMID 16540686
- [Background] Jonkman A, Kaanders JH, Terhaard CH, Hoebers FJ, van den Ende PL, Wijers OB, Verhoef LC, de Jong MA, Leemans CR, Langendijk JA. Multicenter validation of recursive partitioning analysis classification for patients with squamous cell head and neck carcinoma treated with surgery and postoperative radiotherapy. Int J Radiat Oncol Biol Phys. 2007 May 1;68(1):119-25. doi: 10.1016/j.ijrobp.2006.12.002. PMID 17448870
- [Background] Kim T, Giuliano AE, Lyman GH. Lymphatic mapping and sentinel lymph node biopsy in early-stage breast carcinoma: a metaanalysis. Cancer. 2006 Jan 1;106(1):4-16. doi: 10.1002/cncr.21568. PMID 16329134
- [Background] Koller M, Qiu SQ, Linssen MD, Jansen L, Kelder W, de Vries J, Kruithof I, Zhang GJ, Robinson DJ, Nagengast WB, Jorritsma-Smit A, van der Vegt B, van Dam GM. Implementation and benchmarking of a novel analytical framework to clinically evaluate tumor-specific fluorescent tracers. Nat Commun. 2018 Sep 18;9(1):3739. doi: 10.1038/s41467-018-05727-y. PMID 30228269
- [Background] Kumar R, Roy I, Ohulchanskky TY, Vathy LA, Bergey EJ, Sajjad M, Prasad PN. In vivo biodistribution and clearance studies using multimodal organically modified silica nanoparticles. ACS Nano. 2010 Feb 23;4(2):699-708. doi: 10.1021/nn901146y. PMID 20088598
- [Background] Li Y, Zhao T, Wang C, Lin Z, Huang G, Sumer BD, Gao J. Erratum: Molecular basis of cooperativity in pH-triggered supramolecular self-assembly. Nat Commun. 2016 Dec 16;7:13777. doi: 10.1038/ncomms13777. No abstract available. PMID 27981971
- [Background] Ma X, Wang Y, Zhao T, Li Y, Su LC, Wang Z, Huang G, Sumer BD, Gao J. Ultra-pH-sensitive nanoprobe library with broad pH tunability and fluorescence emissions. J Am Chem Soc. 2014 Aug 6;136(31):11085-92. doi: 10.1021/ja5053158. Epub 2014 Jul 29. PMID 25020134
- [Background] Milenovic A, Virag M, Knezevic P, Boras VV, Ostovic KT, Panduric DG, Susic M. Evaluation of sentinel node biopsy in oral carcinomas. Coll Antropol. 2014 Mar;38(1):279-82. PMID 24851630
- [Background] Mo J, Zheng W, Low JJ, Ng J, Ilancheran A, Huang Z. High wavenumber Raman spectroscopy for in vivo detection of cervical dysplasia. Anal Chem. 2009 Nov 1;81(21):8908-15. doi: 10.1021/ac9015159. PMID 19817391
- [Background] Pedersen NJ, Jensen DH, Hedback N, Frendo M, Kiss K, Lelkaitis G, Mortensen J, Christensen A, Specht L, von Buchwald C. Staging of early lymph node metastases with the sentinel lymph node technique and predictive factors in T1/T2 oral cavity cancer: A retrospective single-center study. Head Neck. 2016 Apr;38 Suppl 1:E1033-40. doi: 10.1002/hed.24153. Epub 2015 Sep 2. PMID 26040238
- [Background] Rosenthal EL, Warram JM, de Boer E, Basilion JP, Biel MA, Bogyo M, Bouvet M, Brigman BE, Colson YL, DeMeester SR, Gurtner GC, Ishizawa T, Jacobs PM, Keereweer S, Liao JC, Nguyen QT, Olson JM, Paulsen KD, Rieves D, Sumer BD, Tweedle MF, Vahrmeijer AL, Weichert JP, Wilson BC, Zenn MR, Zinn KR, van Dam GM. Successful Translation of Fluorescence Navigation During Oncologic Surgery: A Consensus Report. J Nucl Med. 2016 Jan;57(1):144-50. doi: 10.2967/jnumed.115.158915. Epub 2015 Oct 8. PMID 26449839
- [Background] Schwarz RA, Gao W, Redden Weber C, Kurachi C, Lee JJ, El-Naggar AK, Richards-Kortum R, Gillenwater AM. Noninvasive evaluation of oral lesions using depth-sensitive optical spectroscopy. Cancer. 2009 Apr 15;115(8):1669-79. doi: 10.1002/cncr.24177. PMID 19170229
- [Background] Sibille M, Patat A, Caplain H, Donazzolo Y. A safety grading scale to support dose escalation and define stopping rules for healthy subject first-entry-into-man studies: some points to consider from the French Club Phase I working group. Br J Clin Pharmacol. 2010 Nov;70(5):736-48. doi: 10.1111/j.1365-2125.2010.03741.x. PMID 21039768
- [Background] Thompson CF, St John MA, Lawson G, Grogan T, Elashoff D, Mendelsohn AH. Diagnostic value of sentinel lymph node biopsy in head and neck cancer: a meta-analysis. Eur Arch Otorhinolaryngol. 2013 Jul;270(7):2115-22. doi: 10.1007/s00405-012-2320-0. Epub 2012 Dec 22. PMID 23263205
- [Background] Vahrmeijer AL, Hutteman M, van der Vorst JR, van de Velde CJ, Frangioni JV. Image-guided cancer surgery using near-infrared fluorescence. Nat Rev Clin Oncol. 2013 Sep;10(9):507-18. doi: 10.1038/nrclinonc.2013.123. Epub 2013 Jul 23. PMID 23881033
- [Background] Wang Y, Zhou K, Huang G, Hensley C, Huang X, Ma X, Zhao T, Sumer BD, DeBerardinis RJ, Gao J. A nanoparticle-based strategy for the imaging of a broad range of tumours by nonlinear amplification of microenvironment signals. Nat Mater. 2014 Feb;13(2):204-12. doi: 10.1038/nmat3819. Epub 2013 Dec 8. PMID 24317187
- [Background] Webb BA, Chimenti M, Jacobson MP, Barber DL. Dysregulated pH: a perfect storm for cancer progression. Nat Rev Cancer. 2011 Aug 11;11(9):671-7. doi: 10.1038/nrc3110. PMID 21833026
- [Background] Zhao T, Huang G, Li Y, Yang S, Ramezani S, Lin Z, Wang Y, Ma X, Zeng Z, Luo M, de Boer E, Xie XJ, Thibodeaux J, Brekken RA, Sun X, Sumer BD, Gao J. A Transistor-like pH Nanoprobe for Tumour Detection and Image-guided Surgery. Nat Biomed Eng. 2016;1:0006. doi: 10.1038/s41551-016-0006. Epub 2016 Dec 19. PMID 28966871
- See also: Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0. National Cancer Institute 27NOV2017 — https://ctep.cancer.gov/protocoldevelopment/
- See also: Declaration of Helsinki — https://www.who.int/publications/journals/bulletin/
- See also: ICH E6 (R2). Integrated addendum to ICH E6(R1): Guideline for good clinical practice. 09NOV2016 — https://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/Efficacy/E6/E6_R2
- See also: FDA Bioanalytical Method Validation Guidance for Industry, May 2018 — http://www.fda.gov/downloads/drugs/guidances/ucm070107.Pdf
- See also: EAFUS - Everything Added to Food in the United States. PEG: ASP, Doc#1285, CAS# 25322-68-3. Polymethacrylate: ASP, Doc# 1406, CAS# 54193-36-1 — https://www.cfsanappsexternal.fda.gov/scripts/fdcc/index.cfm?set=FoodSubstances